CLINICAL TRIAL: NCT03482362
Title: MoTriColor: A Phase II Study of Vinorelbine in Advanced BRAF-like Colon Cancer
Brief Title: Vinorelbine in Advanced BRAF-like Colon Cancer
Acronym: EORTC1616
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Vall d'Hebron Institute of Oncology (Other); Agendia (Industry); European Organisation for Research and Treatment of Cancer - EORTC (Network); Azienda Ospedaliera Niguarda Cà Granda (Other); Fundación para la Investigación del Hospital Clínico de Valencia (Other); University of Campania Luigi Vanvitelli (Other); University of Turin, Italy (Other); Eli Lilly and Company (Industry); Catalan Institute of Health (Other Government); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M16VIB
Record Dates: First submitted 2018-03-13; First posted 2018-03-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2018-08

CONDITIONS: Colon Cancer
Keywords: vinorelbine
MeSH Terms: conditions — Colonic Neoplasms | interventions — Vinorelbine

STUDY DESIGN:
Intervention Model Description: This is a two-stage, single-arm, multi-center, open-label, two-cohort, clinical, phase II, proof of principal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A; KRASmt, BRAFwt, BRAF-like CC (Experimental): Patients with KRAS mutant and BRAF wildtype colon cancer that met the BRAF-like signature according to the validated test of Agendia will be treated with vinorelbine tartrate.
  Interventions: Drug: Vinorelbine Tartrate
- Cohort B; KRASwt, BRAFmt, BRAF-like CC (Experimental): Patients with KRAS wildtype and BRAF mutant colon cancer that met the BRAF-like signature according to the validated test of Agendia will be treated with vinorelbine tartrate.
  Interventions: Drug: Vinorelbine Tartrate

INTERVENTIONS:
Drug: Vinorelbine Tartrate — Intravenous administration of vinorelbine on day 1 and day 8 in a dose of 30 mg/m2. One treatment cycle is 21 days.
  Other Names: Navelbine; Vinorelbine

SUMMARY:
Vecchione et al showed that suppression of RANBP2 results in mitotic defects only in BRAF-like colon cancer (CC) cells, which leads to cell death. Mechanistically, RANBP2 silencing reduces microtubule outgrowth from the kinetochores, thereby inducing spindle perturbations, providing an explanation for the observed mitotic defects. Vinorelbine mimics RANPB2 silencing in BRAF-like and BRAFV600E CC cell lines.

These preclinical data represent a strong rationale to also explore the anti-tumor activity of vinorelbine in patients with advanced BRAF-like (both BRAFm and BRAF wild type) CC. Tumors having this gene signature are referred to as "BRAF-like" and have a similar poor prognosis irrespective of the presence of BRAF(V600E) mutation. Since vinorelbine is standard of care in advanced breast and NSCLC, there is ample experience with the dose and schedule as well as with the safety profile and supportive measures required to prevent side-effects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for this clinical trial (+ TR (translational research)) must be given according to ICH/GCP and national/local regulations
2. Written documentation of BRAF-like signature CC, including BRAFm and BRAFwt, as determined by the validated assay of Agendia
3. Written documentation of KRAS and BRAF mutational status.
4. Age > 18 years
5. Histologically proven and measurable (RECIST criteria v.1.1) metastatic adenocarcinoma of the colon not in a previously irradiated area, treated with at least one or two lines of standard of care therapy, including BRAF inhibitors, for advanced disease
6. WHO performance status of 0-1
7. Able and willing to undergo blood sampling for pharmacodynamic (PD) analysis;
8. Able and willing to undergo tumor biopsy prior to, during and upon treatment;
9. Life expectancy > 3 months allowing adequate follow up of toxicity evaluation and antitumor activity
10. Minimal acceptable safety laboratory values:

    1. ANC > 1.5 x 109 /L
    2. Platelet count > 100 x 109 /L
    3. Hemoglobin > 6.0 mmol/L
    4. Hepatic function as defined by serum bilirubin < 1.5 x ULN, ALAT and ASAT < 2.5 x ULN, or ALAT and ASAT < 5 x ULN in patients with liver metastases
    5. Renal function as defined by serum creatinine < 1.5 x ULN
    6. creatinine clearance > 50 ml/min (by Cockcroft-Gault formula)
11. Negative urine or serum pregnancy test (serum or urine) for female patients with childbearing potential

Exclusion Criteria:

1. Any treatment with investigational drugs, including BRAF inhibitors, within 28 days prior to receiving the first dose of investigational treatment
2. Symptomatic or untreated leptomeningeal disease
3. Symptomatic brain metastasis. Patients previously treated or untreated for these conditions that are asymptomatic in the absence of corticosteroid and anticonvulsant therapy (for at least 4 weeks) are allowed to enroll. Radiotherapy for brain metastasis must have been completed at least 6 weeks prior to start of study treatment. Brain metastasis must be stable with verification by imaging (e.g. brain MRI or CT completed at screening (<21 days before start of treatment) demonstrating no current evidence of progressive brain metastases). Patients are not permitted to receive enzyme inducing anti-epileptic drugs or corticosteroids.
4. Impairment of gastrointestinal (GI) function or GI disease (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, any condition inducing malabsorption, small bowel resection)
5. Other uncontrolled concomitant illness, including serious uncontrolled intercurrent infection
6. Known allergy or any other adverse reaction to any of the drugs or to any related compound
7. Women who are pregnant or breast feeding
8. Unreliable contraceptive methods. Both men and women enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms) 9. Radio-, immuno- or chemotherapy within the last 4 weeks prior to receiving the first dose of investigational treatment. Palliative radiation (1x 8Gy) is allowed

10. Patients who have undergone any major surgery within the last 2 weeks prior to starting study drug or who would not have fully recovered from previous surgery 11. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients 12. Patients with a known history of hepatitis B or C 13. Patients with cardiac comorbidities (myocardial infarct within 6 months of study start, NYHA class ≥ III, congestive heart failure or instable angina pectoris), uncontrolled hypertension (systolic blood pressure > 150 mm Hg and/or diastolic pressure > 90 mm Hg) or prolonged QT-interval (> 440 ms for men, > 460 ms for women) 14. Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for the study 15. Known hypersensitivity to study drug or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Doubling of progression free survival | 15 months
  This means that by vinorelbine treatment the rate of progression drops to 25%.

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 15 months
Overall response rate | 15 months
Duration of response | 15 months
Time to response | 15 months
Overall survival | 15 months
Baseline molecular status (mutation/ expression) in tumor tissue of potential predictive markers of tumor response | 15 months
  The molecular status will be measured by NGS and IHC in tumor tissue.
Gene alterations/expression profiles (i.e. baseline, relapse) in tumor tissue upon progression | 15 months
  The molecular status will be measured by NGS and IHC in tumor tissue.

OTHER OUTCOMES:
Overall response rate of vinorelbine in patients with KRAS mutant, BRAF wildtype, BRAF-like colon cancer vs. KRAS wildtype, BRAF mutant, BRAF-like colon cancer. | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: N Steeghs, MD, PhD, Principal Investigator — NKI-AvL; J Tabernero, Prof, Principal Investigator — VHIO; R Salazar, MD, PhD, Principal Investigator — ICO; R Bernards, Prof, Principal Investigator — Agendia; S Siena, Prof, Principal Investigator — ONCG; A Cervantes, Prof, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA; F Ciardiello, Prof, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA; A Bardelli, Prof, Principal Investigator — UNITO; S Tejpar, Prof, Principal Investigator — UZ Leuven
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: general information — http://www.motricolor.eu